CLINICAL TRIAL: NCT00118495
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Design Trial of the Efficacy and Safety of Zestra(TM) in Women With Mixed Desire/Interest/Arousal/Orgasm Disorders
Brief Title: Zestra in Women With Mixed Sexual Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: QualiLife Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z-04
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Sexual Dysfunction, Psychological
Keywords: female sexual dysfunction; FSD; arousal; orgasm; desire; Zestra; Mixed FSD; Hypoactive sexual desire disorder; Sexual arousal disorder; Orgasmic disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Orgasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Non-prescription Zestra(TM): patented formulation

SUMMARY:
The objective of this study is to evaluate the clinical efficacy and safety of Zestra(TM) in women with acquired mixed desire/interest/arousal/orgasm disorders under conditions of home usage. The primary efficacy hypothesis will compare the effect of Zestra versus placebo on the incidence of "successful and satisfactory" sexual encounters.

DETAILED DESCRIPTION:
This Phase 3 study is being conducted to evaluate the efficacy and safety of Zestra(TM) compared to a placebo oil in women diagnosed as having acquired mixed interest/desire/arousal/orgasm disorders with varying presentations of each component in conditions of home use in conjunction with sexual activities. The study is a randomized, placebo-controlled, double-blind, parallel design trial. After subject screening, there is an open-label, placebo run-in period of four weeks, followed by a double-blinded 12 week treatment period. This design is consistent with the Paris 2003 recommendations for female sexual dysfunction (FSD) clinical trials and the Food and Drug Administration (FDA) Guidance on Clinical Development of Products for the Treatment of Female Sexual Dysfunction although the duration of active treatment in this study is 12 weeks rather than the 6 months suggested by the FDA for Phase 3 studies.

Primary efficacy assessment will be the subjects' assessments of "successful and satisfactory" sexual encounters as recorded in a diary (question 10 in the Female Sexual Encounter Profile [FSEP©]). Secondary evaluations of efficacy will include the other FSEP questions, a subject self-assessment questionnaire (Female Sexual Function Index [FSFI©]), two global assessment questions, a treatment satisfaction questionnaire (WITS©), the Beck Depression Inventory, the Dyadic Adjustment Scale (DAS), a consumer testing survey (QualiLife Consumer Testing Survey [QCTS©]), and a distress scale (Female Sexual Distress Scale [FSDS©]), sexual encounter frequency, and drop-out rates.

The selection of outcome measures in this study is based on the most current information available. The FSEP© has been used in many FSD studies and specifically meets the FDA recommendations for a primary outcome measure. The initial validation study of the FSEP© was presented at the 11th World Congress of the International Society for Sexual and Impotence Research in Buenos Aires in 2004. The FSFI©, the FSDS©, and global assessment questions are routinely used in FSD trials, and the first two have been subjects of ongoing validation for a number of years. Global assessment questions have historically been used to calculate response rates. The QCTS© is a consumer testing survey which addresses issues ultimately impinging on product marketability. WITS© is a female oriented treatment satisfaction instrument newly developed by Stanley E. Althof, Ph.D., Eric W. Corty, Ph.D., and Miki Wieder, M.A., 2004; the authors' authorized use of this instrument in this study is part of the ongoing validation for this questionnaire. Since depression can contribute to FSD and FSD can contribute to depression, seriously confounding diagnostic and treatment schema, the commonly used Beck Depression Inventory will be administered at the end of the baseline run-in period and then at the end of the double-blinded treatment period. Relational factors have the same confounding issues as depression; thus, the participants' attitudes about their relationships with their partners will be assessed at baseline and end of treatment using the Dyadic Adjustment Scale. Sexual encounter frequency may prove a useful outcome measure since a beneficial effect of treatment may be reinforcing, while lack of efficacy by the placebo may be discouraging. A similar hypothesis is the basis of drop-out analysis.

ELIGIBILITY:
Inclusion Criteria:

* Females 21 to 65 years of age.
* Have been previously "functional" or experienced sexual desire/arousal/orgasm for several years in the past.
* Postmenopausal (no menses for one year and appropriate elevation of follicle stimulating hormone [FSH]), or using hormonal contraception for at least 3 months prior to study entry, or have had a tubal ligation at least 3 months prior to study entry or confining all sexual intercourse to a vasectomized partner.
* Provide written informed consent.
* Have a stable heterosexual relationship with a male partner for at least 1 year. Partner must attend screening visit and also sign a separate informed consent form.
* Have a partner score of "not impotent" or "minimally impotent" on the Single Question Assessment of Erectile Dysfunction. The subject will determine the partner score privately.
* Willing to engage in sexual activities with intent to attain orgasm at least 2 times per week.
* Meet the diagnostic criteria for one or more of the following acquired disorders:

  * Women's sexual interest/desire disorder;
  * Subjective sexual arousal disorder;
  * Combined genital and subjective arousal disorder;
  * Genital sexual arousal disorder;
  * Women's orgasmic disorder.
* Have a score of > 15 on the FSDS .
* Willing and able to understand and comply with all study requirements.

Exclusion Criteria:

* Evidence of unresolved sexual trauma or abuse.
* Primary anorgasmia, vaginismus, sexual pain disorder, sexual aversion disorder, or persistent sexual arousal disorder.
* Female sexual dysfunction caused by untreated endocrine disease, e.g., hypopituitarism, hypothyroidism, diabetes mellitus.
* Pregnant or nursing.
* Sensitivity to any of the ingredients in Zestra for Women(TM).
* Chronic or complicated urinary tract or vaginal infections within previous 12 months.
* Pelvic inflammatory disease within previous 12 months.
* Currently active sexually transmitted disease.
* Chronic dyspareunia not attributable to vaginal dryness within previous 12 months.
* Currently active moderate to severe vaginitis.
* Cervical dysplasia within previous 12 months.
* Significant cervicitis as manifested by mucopurulent discharge from the cervix.
* Significant gynecologic conditions such as uterine fibroids, vulvar vestibulitis, or vaginismus that may (in the investigator's opinion) interfere with the subject's ability to comply with study procedures.
* Psychoses and bipolar disorder.
* Use of neuroleptics or lithium within previous 3 months.
* Unwillingness to forego any medications, herbal treatments, or dietary supplements intended to enhance sexual function during the course of the study.
* History of myocardial infarction within previous 6 months.
* History or evidence of significant renal or hepatic disease within previous 6 months.
* Significant central nervous system diseases within the last 6 months, i.e., stroke, spinal cord injury, multiple sclerosis, etc.
* Unwillingness to omit cunnilingus from sexual activities during the study. No post-coital fellatio allowed.
* Any condition which, in the Investigator's opinion, would interfere with the subject's ability to provide informed consent, to comply with study instructions, or which might confound the interpretation of the study results.
* Any condition which would endanger the participant if she participated in this trial.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Safety: adverse events, physical examinations, clinical laboratory evaluations
Female Sexual Function Index domain scores and totals | Baseline to Visit 6 (12 weeks)

SECONDARY OUTCOMES:
Efficacy: incidences for remaining FSEP© questions, FSFI© (all domains), FSDS©, global assessment questions, WITS©, QCTS©, Beck Depression Inventory, Dyadic Adjustment Scale, sexual encounter frequency, drop out rates

CONTACTS AND LOCATIONS:
Overall Officials: David M Ferguson, PhD, MD, FACCP, Study Director — Clinical Research Services Consulting; Julia R Heiman, PhD, Principal Investigator — Kinsey Institute for Research in Sex, Gender and Reproduction
Locations (13):
- United States (13):
  - West Coast Clinical Research, Tarzana, California
  - Urology Research Options, Aurora, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Center for Marital and Sexual Health of South Florida, West Palm Beach, Florida
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Outpatient Clinical Research Facility, Indianapolis, Indiana
  - Lahey Clinic, Peabody, Massachusetts
  - Accumed Research Associates, Garden City, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Pelvic and Sexual Health Institute, Philadelphia, Pennsylvania
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Midwest Research Specialists, LLC, Milwaukee, Wisconsin

REFERENCES:
- [Background] Ferguson DM, Steidle CP, Singh GS, Alexander JS, Weihmiller MK, Crosby MG. Randomized, placebo-controlled, double blind, crossover design trial of the efficacy and safety of Zestra for Women in women with and without female sexual arousal disorder. J Sex Marital Ther. 2003;29 Suppl 1:33-44. doi: 10.1080/713847125. PMID 12735087